CLINICAL TRIAL: NCT04031157
Title: A Prospective, Randomized, Controlled Study to Evaluate the Safety and Efficacy of the Predictix Antidepressant Clinician Support Tool in Prescribing Antidepressant Medication for the Treatment of Patients Diagnosed With Major Depressive Disorder
Brief Title: Controlled Study to Evaluate the Safety and Efficacy of the Predictix Antidepressant Clinician Support Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taliaz Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CL-02-PRT-02
Record Dates: First submitted 2019-07-14; First posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGT arm (Experimental): Predictix Antidepressant-guided treatment condition
  Interventions: Device: Predictix Antidepressant
- soc arm (No Intervention): Standard of Care condition

INTERVENTIONS:
Device: Predictix Antidepressant — Predictix Antidepressant guided treatment
  Arms: PGT arm

SUMMARY:
The study will compare two groups of patients: a control group of patients treated per the Standard of Care when prescribed with a medication for their Major depression disorder, versus a group of patients that used the Predictix Antidepressant tool when prescribed with a medication for their Major depression disorder by their treating physician. Success will be measured by the number (proportion) of responders per group.

DETAILED DESCRIPTION:
The study will be comprised of two arms:

1. PGT arm - Predictix Antidepressant-guided treatment condition
2. SOC (control) arm - Standard of Care condition Eligible subjects will be assigned to one of the study arms at a 1:1 ratio and will be followed for a period of 12 weeks.

An assigned psychiatric expert will review and approve subject's eligibility prior to entrance to the study, as well as, the medication/s prescribed based on the Predictix report prior to treatment start.

During the 12 weeks of follow up , data will be collected at the following timepoints: Screening, Baseline (start of treatment) and at 4, 8 and 12 weeks.

Visits will include the completion of several questionnaires designed to answer the study objectives, either as self-reported by the patients and/ or by the physician.

Depression scores by the Quick Inventory of Depressive Symptomatology (QIDS 16) questionnaire and evaluation of all safety related endpoints will be analyzed following the completion of the 12 weeks visit procedures. In case of a change in treatment, as per the treating physician's decision, a new 12 weeks cycle of data collection will start. Two independent cycles are permitted per patient.

In addition, retrospective (6 months prior to enrollment) and long-term follow up period data (12 months post enrollment) will be analyzed, in order to evaluate the device use effect on patients care outcomes in terms of economic burden and Social impact, on patients, employers, the health care system and payers.

The analysis will be based on both the work productivity and activity impairment questionnaire and the patient's electronic medical data record.

ELIGIBILITY:
Inclusion Criteria:

* Male and female at the age of 18 - 75 years old at time of screening.
* MDD diagnosis per DSM V at screening visit or prior to screening visit.
* Rule out other causes of depressive symptoms other than MDD.
* Ability to read, understand and sign an informed consent document
* Female subjects at reproductive age that are tested negative for pregnancy
* Women with childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods during the whole study duration

Exclusion Criteria:

* Patient is currently on an antidepressant treatment.
* Patient is diagnosed with other major psychopathologies (i.e. schizophrenia, bipolar disorder, psychotic depression, geriatric depression).
* requires antipsychotic medication or mood stabilizers.
* Patient is at substantial suicidal risk as judged by the treating physician
* Patient has attempted suicide in the past year.
* Patient has any current unstable medical condition or surgical illness.
* Patient has history of seizure or convulsions.
* Patient has history of drug abuse or alcoholism in the last 6 months.
* Inadequate communication with the patient.
* Patient has participated in another clinical study in the last 30 days preceding this study.
* In the investigator's judgement, patient is not able to provide written informed consent and follow protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate in the PGT and SOC groups | 12 weeks
  Overall Response rate with and without the use of the Predictix Antidepressant software tool. Response is measures as at least 45% reduction in symptoms severity, measured by the Quick Inventory of Depressive Symptomatology (QIDS 16)

SECONDARY OUTCOMES:
Change from baseline in Quick Inventory of Depressive Symptomatology( QIDS 16) self reported score | 12 weeks
  Change in total score of the self reported questionnaire. Total score range is 0-48
Usability and satisfaction of the Predictix tool | 12 weeks
  review of completed questionnaires by the treating family physician/general practitioner and psychiatric expert. Total score rate in 12-84. (higher value represent better outcome)
Economic burden* and social impact on patients, employers, the health system and payers | 12 month
  Based on the analysis of the patients' electronic medical data record retrospectively (6 months prior to enrollment) and following a long-term follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi healthcare services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No